CLINICAL TRIAL: NCT04348630
Title: Health Canada - Establishing Evidence-based Indoor Temperature Thresholds to Protect Health
Brief Title: Establishing Evidence-based Indoor Temperature Thresholds to Protect Health
Acronym: HW2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Glen P. Kenny, Full Professor, University Research Chair, University of Ottawa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2018-026H
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Aging; Heat Stress; Physiological Stress
Keywords: Heatwave,; heat-vulnerability; Indoor environments; Cardiovascular strain; thermoregulation; heat strain
MeSH Terms: conditions — Heat Stress Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participant identifier and experimental arm will be blinded from investigator responsible for analyzing outcomes in the cardiovascular battery (see detailed description).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HOT condition (Experimental): Participants are exposed to 36°C and 45% relative humidity for 8 hours. These conditions were chosen to represent an extreme heat condition (i.e., heatwave) and are similar to peak domicile conditions measured in low-income high-rise apartment complexes during heatwaves.
  Interventions: Other: Simulated heatwave exposure
- WARM Condition (Experimental): Participants are exposed to 31°C and 45% relative humidity for 8 hours. These conditions are similar to mean domicile conditions measured in a variety of domicile types during heat waves complexes during heatwaves and are consistent with the World Heath Organization recommendation for maximal indoor temperatures.
  Interventions: Other: Simulated heatwave exposure
- TEMPERATE Condition (Experimental): Participants are exposed to 26°C and 45% relative humidity for 8 hours. These conditions are consistent with Toronto Public Health recommendation for maximal indoor temperatures, which are based on the increase in mortality associated with increases in outdoor temperature above these limits.
  Interventions: Other: Simulated heatwave exposure
- COOL Condition (Experimental): Participants are exposed to 22°C and 45% relative humidity for 8 hours. These conditions are consistent with actively cooled (air-conditioned) domicile.
  Interventions: Other: Simulated heatwave exposure

INTERVENTIONS:
Other: Simulated heatwave exposure — Older adults are exposed to a 8-hour simulated exposure

SUMMARY:
An individual's ability to adequately cope with short- or long-term increases in ambient temperature is critical for maintaining health and wellbeing. Prolonged increases in temperature (heatwaves) pose a serious health risk for older adults, who have a reduced capacity to regulate body temperature. Currently, however, there is a lack of information regarding how different environmental conditions experienced during heatwaves impact body temperature regulation and physiological function. This is particularly important in the context of ambient conditions in the home, where older adults spend the majority of their time. This project will address this important issue by exposing healthy older adults to prolonged (8-hour) simulated heatwaves comprising a range of environmental conditions representative of an actively cooled domicile through to a worst-case scenario (i.e., no capacity for home cooling). The investigators will directly measure their ability to regulate their body temperature and the associated impact on the autonomic control of the heart. The investigators anticipate that physiological strain will be mild during prolonged exposure to conditions below the currently recommended thresholds set by Toronto Public Health (26°C). However, at higher indoor temperatures, impairments in body temperature and cardiovascular regulation will be seen.

DETAILED DESCRIPTION:
OBJECTIVES

The objective of this project is to evaluate the effect of a range of environments experienced during heatwaves on body temperature and autonomic cardiovascular function in older adults. This will be accomplished by comparing thermal and cardiovascular responses in a group of older adults resting for 8-hours in a range of conditions representative of those experienced indoors during heatwaves. To assess how the strain experienced in these conditions affects haemodynamic regulation in turn, this study will also include validated tests of cardiovascular autonomic function.

Hypotheses

Indices of thermal and cardiovascular strain will not be appreciably modified in older adults resting in simulated indoor environments below the currently recommended thresholds set by Toronto Public Health (22°C and 26°C). However, at higher indoor temperatures (31°C and 36°C) thermal and cardiovascular responses will be elevated. The increased physiological strain in these conditions will be reflected in attenuated responses to validated cardiovascular autonomic functional tests.

METHODS

Participants A total of 16 older (age: 65-80 years) adults will be recruited for the proposed project with an approximately even distribution of men and women. Each participant will complete each of the 4 experimental arms of the study. Recruited participants will be homogeneous for anthropomorphic characteristics and as well as habitual physical activity levels as verified via standardized questionnaires (determined during a preliminary session). Written and informed consent will be obtained from all volunteers prior to participation.

Study Design

Pre-trial instructions

All participants will be asked to avoid strenuous activity and alcohol for 24 hours prior to all preliminary and experimental sessions and to eat a light meal 2 hours before the start of each session. Participants will also be asked to consume a minimum of 500 ml of water the night before and morning of each session to ensure adequate hydration. Adequate hydration will be verified upon arrival to the laboratory via urine specific gravity (urine specific gravity <1.025). Participants will wear an athletic top and shorts for all sessions.

Preliminary screening

All participants will complete one preliminary evaluation a minimum of 48 hours before the first experimental session. During this session they will be familiarized with all experimental procedures and measurement techniques and will complete the Get Active Questionnaire (GAQ) and the American Heart Association Pre-participation screening Questionnaire to assess their eligibility to participate. The GAQ will also be used to assess habitual activity levels along with the Kohl Physical Activity Questionnaire. Participants will also provide verbal and written informed consent at this time. Thereafter, participant physical characteristics will be evaluated. Body height and mass will be determined via a physician stadiometer and a high-performance weighing terminal, respectively, and from these measurements body surface area will be calculated. Body density will be estimated via hydrostatic weighing and used to calculate body fat percentage.

Experimental Protocol Each experimental session will commence at approximately 08:00. Upon arrival to the laboratory the participant will provide a urine sample for measurement of urine specific gravity and insert a rectal temperature probe. Thereafter, participants will be instrumented for the measurement of skin temperature. A measurement of body mass (nude) will also be taken at this time. Participants will then be transferred to a thermal chamber regulated to 22°C and 45%. Following 10-min of supine rest, participants will perform a specialized cardiovascular test battery (see below). They will then rest in the seated position in a room immediately adjacent to the thermal (~22°C) chamber for ~30 min while baseline body temperatures and cardiovascular measures are recorded. A venous blood sample will be obtained at this time.

While baseline measurements are being taken, the thermal chamber will be heated to the conditions for that day's session. Each participant will complete four separate sessions consisting of resting exposure to: i) 36°C, based on maximal measured indoor temperatures (i.e., 35°C) and similar to outdoor conditions experienced during recent heatwaves in North America (HOT); ii) 31°C, similar average daytime temperature during the 2010 heatwave in Ontario and Quebec as well as the World Health Organization recommended indoor temperature limit during heatwaves (WARM); iii) 26°C corresponding to recommended upper limits for indoor environments as set by Toronto Public Health (TEMPERATE) and iv) 22°C, to simulate an air-conditioned environment (COOL). In all sessions, relative humidity will be set to 45%.

Following baseline, the participant will enter the thermal chamber where they will rest for 8 hours. They will spend the majority of this time in the seated (slightly reclined) position, except for at the 6th hour where they will again perform the cardiovascular test battery. Rectal and skin temperatures and heart rate will be measured continuously throughout exposure. Tap water will be provided ad libitum from a ~500 mL cup placed on a side-table positioned slightly behind the participant. Participants will also be allowed to eat a self-provided lunch between hours 1.5 and 3.5 of exposure. Every 60 min, arterial blood pressure and heart rate will be measured in triplicate after which participants will stand to provide a measurement of body mass in order to determine sweat losses. At this time. participants will be allowed to remain standing and briefly perform light stretching, if desired (max ~5 min).

Autonomic control of heart rate and blood pressure will be assessed prior to and at the end of each session using a battery of cardiovascular tests, which, in Study B consists of: i) analysis of heart rate variability and spontaneous baroreflex sensitivity during supine rest, ii) Ewing's battery (modified) for assessment of cardiovascular autonomic function, and iii) analysis of integrated baroreflex sensitivity during cyclical perturbations in arterial pressure evoked by stand-squat maneuvers. Prior to the battery, participants will be instrumented with an integrated 3-lead ECG non-invasive blood pressure monitor for the integrated measurement of beat-to-beat heart rate and arterial blood pressure, estimated from the arterial pressure waveform measured at the left middle finger. The same researcher will administer the battery for all sessions. Finally, note that the first two sections of the battery described below will be performed twice in succession prior to the stand-squat procedures.

Following 8-min of supine rest, heart rate variability (HRV) and baroreflex sensitivity (BRS) will be evaluated during 8-min of supine rest. Participants will be instructed to breathe (diaphragmatic) in time with a metronome set to 30 beats/min, to remove the influence of respiratory sinus rhythm on cyclical fluctuations in heart rate and blood pressure. Thereafter, the metronome will be stopped and 1-min of recovery will be given prior to the start of the Ewing's battery.

The modified Ewing's battery to be employed consists of three tests designed to assess autonomic control of heart rate and blood pressure. First, participants perform 1 min of deep diaphragmatic breathing at a rate of 6 breaths/min. Breathing will be performed to vital capacity - that is, through a maximal inspiration and expiration. 5-min of recovery will be given before the next test. The next test is the Valsalva maneuver. While still in the supine position, participants will exhale against a closed glottis into a narrow vinyl tube connected to an electronic pressure transducer that will be used to provide constant feedback to the participant on the generated expiratory pressure. The participant will be instructed to maintain a constant pressure of 40 mmHg for 15 s. Throughout expiratory straining, air will be vented via a small bleed to prevent generation pressure via the mouth. Upon release, heart rate and blood pressure will be monitored for 1 min. The final test is the lying-to-standing test. Following 1-min of rest in the supine position, the participant is instructed to quickly assume a standing position directly beside the bed. The participant then stands quietly for 3 min while heart rate and blood pressure are monitored.

Following the second Ewing's battery, the participant will rest in the seated position on a rigid chair for 10 mins. The participant will then be asked to stand for 90-seconds while the positioning of the sling and finger-pressure cuff is adjusted (if needed) to ensure the left hand is maintained at heart-level. After this, 5-min of squat-stands will be performed at a rate of 6 cycles/min. Each cycle will consist of a squat, held for 5 seconds, followed by standing for 5 sec. For these maneuvers, participants will be instructed to maintain a consistent depth for each squat, breath normally to avoid expiratory straining and limit excessive forward flexion at the hip.

After the cardiovascular battery, participants will remain seated in the chamber for the remainder of the 8-hour exposure (~45 min). Following measurements of arterial blood pressure, a final venous blood sample will be obtained followed by a measurement of body mass. The participant will be provided with water and/or a commercially available sports drink before leaving laboratory.

Data analysis

Continuous variables related to thermal strain and cardiovascular strain will be converted to 15-min averages for baseline and at each hour of exposure. Likewise, seated arterial pressures (3 measurement average) will be presented at these time points. Rate pressure product will be calculated as the product of heart rate and systolic blood pressure. The change in body mass from baseline values will also be determined at each hour of exposure to quantify the rate of fluid loss, corrected for fluid consumed and urination. The change in plasma volume and serum osmolality from baseline to end exposure will also be calculated from the venous blood samples obtained at the start and end of each session. HRV and resting spontaneous cardiac BRS will be determined from data collected during the 8-min controlled breathing period. Similarly, integrated BRS will be derived from collected blood pressure and ECG waveforms collected during the stand-squat maneuvers.

For the clinically validated tests in the Ewing battery, analysis will be performed by a trained researcher blinded to the participant and session code (i.e., environmental conditions). Deep breathing will be analysed as the difference in heart rate between the average of the three lowest and three highest values recorded during inspiration and expiration, respectively (E/I HRDiff). For the Valsalva maneuver, the so-called Valsalva ratio (VALratio) is calculated as the longest R-R interval during recovery divided by the shortest R-R interval during straining. Finally, the lying to standing test is analysed by determination of the 30:15 ratio, which represents the longest RR interval measured between the 25-35th heart beat upon standing divided by the shortest RR interval between the 10-20th beat after standing. Additionally, the systolic response to standing (SRstand) is also taken as the 1-min average of systolic blood pressure after the second min of standing divided by systolic blood pressure during the pre-stand supine resting period (i.e., the reduction in systolic pressure upon assuming a standing position). Values for each test will be taken as the average of each of the two recorded values.

Statistical analysis and sample size calculation

Statistical analysis will compare end-exposure data relating to thermal and cardiovascular strain as well as autonomic function (while correcting for between-session baseline variability). Body temperature and cardiovascular responses at the end of exposure (i.e., hour 8) as well as the autonomic functional tests of the cardiovascular battery will be evaluated using an analysis of covariance (ANCOVA) with the repeated factor of environmental condition and baseline values modeled as a continuous covariate. Variables related to fluid loss (e.g., change in body mass, plasma volume and serum osmolality) will be analysed via a one-way ANOVA with the factor of condition (4 levels). For all statistical models, homogeneity of variances will be assessed using Levene's test. Normal distribution of residuals will be assessed with Sharpiro-Wilks test and visual inspection of histograms and Q-Q plots and data will be log-transformed in the event that distribution of residuals deviates from normality. Pre-planned post hoc comparisons will be employed to identify differences between adjacent conditions (e.g., COOL vs TEMP, TEMP vs. WARM, WARM vs. HOT) in order to limit a large family of comparisons. For all analyses, alpha will be set at P < 0.050. Descriptive statistics will be presented as mean (standard deviation). Comparisons between groups or time-points (where appropriate) will be presented as means ± 95% confidence interval.

An a priori power analysis determined that a total sample size of 16 older adults is required to detect a difference in rectal temperature between groups with 80% statistical power, after adjusting for multiple comparisons. The effect size (Cohen's d=1.0) was determined based on practically meaningful difference of 0.3°C between conditions, assuming a standard deviation of 0.3. The standard deviation was based on previously published studies from our laboratory, which demonstrated a 0.2°C (SD 0.3) difference in core temperature between young and older adults and a 0.0°C (SD 0.3) difference in core temperature between older adults with and without type 2 diabetes following 3 hours of rest in a hot environment (40°C, 30% relative humidity).

ELIGIBILITY:
Inclusion Criteria:

* Male or female (non-pregnant) adults aged 18-80 with or without a) chronic hypertension (elevated resting blood pressure; as defined by Heart and Stroke Canada and Hypertension Canada), b) type 2 diabetes as defined by Diabetes Canada, with at least 5 years having elapsed since time of diagnosis and or c) obesity as defined by the World Health Organization (Body Mass Index [BMI] greater than or equal to 30)
* non-smoking.

Exclusion Criteria:

- Episode(s) of severe hypoglycemia (requiring the assistance of another person) within the previous year, or inability to sense hypoglycemia (hypoglycemia unawareness).

Serious complications related to your diabetes (gastroparesis, renal disease, uncontrolled hypertension, severe autonomic neuropathy).

* Uncontrolled hypertension - BP >150 mmHg systolic or >95 mmHg diastolic in a sitting position.
* Restrictions in physical activity due to disease (e.g. intermittent claudication, renal impairment, active proliferative retinopathy, unstable cardiac or pulmonary disease, disabling stroke, severe arthritis, etc.).
* Use of or changes in medication judged by the patient or investigators to make participation in this study inadvisable.
* Cardiac abnormalities identified in your physical health screening form (adults <65 years of age and older; adults <60 years of age and older with diabetes and or hypertension) or during exercise stress testing as assessed by 12-lead (all adults ≥65 years of age and older).

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Rectal temperature | Final 15 min of exposures
  Index of core body temperature
Mean skin temperature | Final 15 min of exposures
  Calculated based on skin temperature measured over 8 body regions

SECONDARY OUTCOMES:
Heart rate | Final 15 min of exposures
  Measured continuously throughout exposure
Arterial blood pressures | Final 15 min of exposures
  Systolic pressure, diastolic pressure, mean arterial pressure
Rate pressure product | Final 15 min of exposures
  Calculated as systolic blood pressure multiplied by heart rate
Ewings battery tests | Hour 6 of exposure
  Deep breathing, valsalva maneuver, 30:15 ratio, systolic response to standing
Resting heart rate variability | Hour 6 of exposure
  Derived from data collected during supine rest with controlled breathing
Resting cardiac baroreflex sensitivity | Hour 6 of exposure
  Derived from data collected during supine rest with controlled breathing
Integrated baroreflex sensitivity | Hour 6 of exposure
  Derived from data collected during stand-squat procedures
Change in body weight | Hour 8 of exposure
  Surrogate of fluid loss
Change in plasma volume | Hour 8 of exposure
  Determined from venous blood samples
Serum osmolality | Hour 8 of exposure
  Determined from venous blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Glen P Kenny, PhD, Principal Investigator — University of Ottawa; Ronald J Sigal, MD, MPH, Principal Investigator — University of Calgary
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT04348630/Prot_SAP_000.pdf